CLINICAL TRIAL: NCT03688477
Title: A Post-Market, Prospective Study to Evaluate the Iovera° Device in Treating Pain Associated With Anterior Cruciate Ligament Reconstruction and Rehabilitation
Brief Title: Iovera° to Treat Pain Associated With ACL Reconstruction and Rehabilitation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting patients
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MYO-1348
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iovera° (Experimental): Patients will receive iovera° prior to stand of care ACL
  Interventions: Device: iovera°
- Standard of Care (No Intervention): Patients will receive standard of care ACL procedure without iovera° treatment.

INTERVENTIONS:
Device: iovera° — iovera° is minimally-invasive procedure using cold to target sensory nerve tissue and provide temporary pain relief through cryoneurolysis. The iovera° device uses well-established principles of cryobiology to temporarily deactivate sensory nerves that contribute to pain
  Arms: iovera°

SUMMARY:
To evaluate the outcomes of patients undergoing iovera° treatment of the ISN and AFCN on postoperative knee pain and function following anterior cruciate ligament reconstruction

DETAILED DESCRIPTION:
The most commonly reconstructed ligament in the knee is the anterior cruciate ligament (ACL)1. In 2006 a total of 134,421 ACL reconstructions were performed in the United States, representing a 37% increase in procedures since 19941. Today, most ACL reconstructions are performed on an outpatient basis2. While this has led to improvements in patient satisfaction3 and cost4, it has simultaneously resulted in more complicated postoperative pain management. Managing this pain via multi-modal strategies, including peripheral nerve blocks, in the postoperative phase has been shown to decrease opioid related side effects, decrease hospital stay, and increase time to ambulation5. Nursing, hospital, and pharmacy utilization in managing PCA, continuous regional nerve blocks, and administration of oral opioid dosing are associated with higher costs of care and introduce sources for staff error6,7. Furthermore, the idea of multi-modal pain management extends beyond the surgical procedure. Decreasing prescription opioid use during outpatient rehabilitation decreases NSAID and opioid related side effects8.

Myoscience, Inc. (Fremont, CA) has developed a device - iovera° - as a novel, minimally-invasive procedure using cold to target sensory nerve tissue and provide temporary pain relief through cryoneurolysis. The iovera° device uses well-established principles of cryobiology to temporarily deactivate sensory nerves that contribute to pain. Prior studies of the iovera° device have provided evidence of effectiveness and safety for treatment of the Infrapatellar Branch of the Saphenous Nerve and another study has demonstrated that a short-term block of this nerve resulted in reduced pain following an ACL repair.9

In a multicenter, double-blind, sham-controlled, randomized trial sponsored by Myoscience, Inc, the iovera° device was shown to temporarily relieve pain in patients with osteoarthritis of the knee. Compared to the sham group, patients who received active treatment had a statistically significant greater change from baseline in the WOMAC pain subscale score at Day 30 (p=0.0004), Day 60 (p=0.0176), and Day 90 (p=0.0061). Patients deemed WOMAC pain responders at Day 120 continued to experience a statistically significant treatment effect at Day 150. Most expected side effects were mild in severity and resolved within 30 days. The incidence of device- or procedure-related adverse events was similar in the two treatment groups with no occurrence of serious or unanticipated adverse events.10

The goal of the study described herein is to determine the safety and efficacy of the iovera° treatment for reducing the pain associated with anterior cruciate ligament (ACL) reconstruction and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 49 years of age
2. Scheduled to undergo unilateral anterior cruciate ligament reconstruction with patellar tendon autograft
3. In the opinion of the investigator, the subject is an active participant in recreational or competitive sports, physical activity, or other fitness regimen at the time of ACL injury and is seeking repair to help return to sport or activity
4. Subject is willing and able to give written informed consent.
5. Subject is fluent in verbal and written English.
6. Subject is willing and able to comply with study instructions and commit to all follow-up visits for the duration of the study.
7. Subject is in good general health and free of any systemic disease state or physical condition that might impair evaluation or which in the Investigator's opinion, exposes the Subject to an unacceptable risk by study participation.

Exclusion Criteria:

1. Prior ligamentous injury and/or surgery of either knee (arthroscopic surgeries allowed), contralateral ACL reconstruction, previous ACL surgery of the target knee, previous graft failure, or relevant musculoskeletal impairment
2. Prior surgery or injury in the knee or treatment areas that may have altered the anatomy of the target nerves or resulted in scar tissue in the iovera° treatment areas.
3. Any pain disorder, neuro-muscular disorder, or neuropathy that in the opinion of the Investigator may confound post-operative assessments for pain or rehabilitation. Examples include but are not limited to: fibromyalgia, diabetic neuropathy, multiple sclerosis, etc.
4. History of opioid or alcohol abuse within past 3 years.
5. Open and/or infected wound in the treatment areas or any local skin condition at the treatment sites that in the Investigator's opinion would adversely affect treatment or outcomes.
6. History of cryoglobulinemia
7. History of paroxysmal cold hemoglobinuria.
8. History of cold urticaria.
9. History of Raynaud's disease.
10. Any chronic medical condition that in the Investigator's opinion would prevent adequate participation.
11. Any chronic medication use (prescription, over-the-counter, etc.) that in the Investigator's opinion would affect study participation or Subject safety.
12. For any reason, in the opinion of the Investigator, the Subject may not be a suitable candidate for study participation (i.e., worker's compensation, history of noncompliance, drug dependency, etc.).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Cumulative Opioid Consumption | 3 months
  The number of opioid pills consumed over a 6 week period following TKA surgery. The amount of pills consumed is determined based on a count of remaining pills that occurs at each follow-up versus the amount dispensed to the subject.

SECONDARY OUTCOMES:
Numerical Rating Score (NRS) for Pain | 3 months
  The NRS is an 11-point scale (0 points to 10 points), where 0 points equals "no pain" and 10 points equals the "worst pain".
International Knee Documentation Committee (IKDC) Score | 3 months
  The International Knee Documentation Committee (IKDC Questionnaire) is a knee-specific patient-reported outcome measure. IKDC has been subjected to rigorous statistical evaluation and has proven to be a valid and responsive patient-reported outcome measure. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. Scores are obtained by summing the individual items, then transforming the crude total to a scaled number that ranges from 0 to 100. This final number is interpreted as a measure of function with higher scores representing higher levels of function.
Active Range of Motion - Extension and Flexion | 3 months
  Movement Extension: Have the participant lie in a supine position on an examining table with the head of the table elevated to about 25 to 30 degrees. The leg measured should be extended. The participant should tighten their quadriceps muscles to actively extend their knee (push their knee into the table) three times. On the third trial, the Investigator or Designee measures the angle in degrees using the goniometer.
  Movement Flexion: After the knee extension measurement is taken the bolster is removed and the participant is asked to place their foot as close as possible to their buttocks (foot on the table). After the knee flexion measurement is taken (on the third trial), the participant is told that they can extend their leg and relax. Examiner measures the angle in degrees using the goniometer.
Straight Leg Raise | 3 months
  The straight leg raise immediately after surgery can be completed with the use of a knee brace at the investigator's discretion.
  To perform this initial straight leg raise, the subject will lie supine, bend the unaffected knee, and keep the surgical knee straight. The subject will attempt to contract their quadriceps by straightening the surgical knee all the way, and slowly lift their leg up off the floor. The subject should try to lift their legs to a maximum of 12 inches, hold it in this position for one or two seconds, and then slowly lower their leg down. This exercise should be repeated until subject failure or to a maximum of 20 repetitions.
  The number of repetitions will be recorded in subject source. If no repetitions are completed, the score is 0. If the subject displays an extension lag and cannot straighten their leg despite being able to raise it, the score is 0.

CONTACTS AND LOCATIONS:
Locations (1):
- SurgiCare of Manhattan, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided